CLINICAL TRIAL: NCT02036905
Title: Comparing the Early Use of Cervical/Upper Thoracic Mobilization and Manipulation for Individuals With Mechanical Neck Pain.
Brief Title: Cervical and Upper Thoracic Mobilization and Manipulation for Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Collaborators: Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Kenneth Learman, Dr. Kenneth Learman, Youngstown State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 181-13
Record Dates: First submitted 2013-07-15; First posted 2014-01-15 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Neck Pain
Keywords: neck pain, orthopedic manual therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical and thoracic mobilization (Experimental): Cervical and thoracic mobilization: described as a repetitive low-velocity oscillatory movement applied to a joint segment. It is graded 1-4 based on the size of the amplitude and where in range it is being applied. The mobilization technique chosen will be based on the examination and clinical reasoning process of the therapist. The cervical and thoracic mobilization will be applied to the most provocative level.
  Interventions: Other: Cervical and thoracic mobilization
- Cervical and thoracic manipulation (Experimental): Cervical and thoracic manipulation: is defined as high-velocity low-amplitude thrust at end range of a particular spinal segment. The therapist performs this technique by taking up all available slack at a particular segment and applying a high-velocity thrust through the end-range restriction. The manipulation technique will be chosen based on the examination and clinical reasoning process of the therapist.
  Interventions: Other: cervical and thoracic manipulation

INTERVENTIONS:
Other: Cervical and thoracic mobilization — Described in arm description
  Arms: Cervical and thoracic mobilization
Other: cervical and thoracic manipulation — described in arm description
  Arms: Cervical and thoracic manipulation

SUMMARY:
The objective of this pilot study is to determine the feasibility of a large-scale trial. The primary objective is to determine if manipulation applied to the cervical and thoracic spines is more effective than mobilization applied to the cervical and thoracic spines for the management of patients with mechanical neck pain.

DETAILED DESCRIPTION:
All potential subjects will be assessed for eligibility prior to signing the informed consent by filling out a demographic questionnaire and through a subjective interview that will include a health history examination performed by a physical therapist that has received additional training in orthopedic manual therapy. A physical therapist (PT) is a highly educated licensed health care professional that has graduated from an accredited university and has passed a national licensure exam. Physical therapists specialize in movement disorders and are well trained in the examination and treatment for primary and secondary medical conditions pertaining to the cardiovascular, neuromuscular, musculoskeletal, and integumentary body systems. Manual therapy interventions for the neck and thoracic spine including manipulations are taught in entry-level physical therapy programs. Continuing education courses are available for physical therapists to get advanced training in manual therapy. This training involves not only improving the skill set of the therapist but also focuses on enhancing the knowledge of the therapist concerning the safety of patients. Each of the treating therapists will have certifications in manual therapy. Screening for inclusion and exclusion criteria will be done by the treating PT by means of assessing subjective outcomes, patient demographic, and through their subjective history examine. Subjects will then be given the informed consent to be read and signed if they agree to participate. Subjects will be permitted to ask any questions relative to any study procedures they do not understand. Two physical therapists at each facility will be used in order to keep the outcome measures blinded. The treating therapist or clinic PT will perform the examination/evaluation and perform all manual therapy treatments during the first 2 visits of care. Pending there are no scheduling conflicts; the treating therapist will continue to provide the treatment. If there is a scheduling conflict, another physical therapist will provide the patient's care until the next available opening on the treating therapist. The recording therapist, or research therapist, will record all the dependent variables and will remain blinded to group allocation. This is the only assignment given to the research therapist. The treating therapist will be blinded to all results of the outcome data except in the case where data is needed for clinical decision making in order to optimize patient outcomes. After informed consent is attained, outcome data will then be collected by the recording physical therapist that is not aware of group allocation. The data collected will include the neck disability index (NDI), patient specific functional score (PSFS), numeric pain rating scale (NPRS), deep cervical flexion test (DCF), cervical range of motion (CROM) using a CROM, therapist equipoise, and patient preference. Following initial data collection, each subject will be randomized via concealed allocation to receive either mobilization or manipulation directed to the cervical and upper thoracic spine for the first two treatment visits. The patient will be treated on day 1 with their randomized treatment technique. The manual technique chosen for treatment by each clinician will be determined by the results of their physical examination. Other interventions included for both groups will include a standardized exercise program and advice, encouragement, and assurance. Immediately following the treatment procedures, data will be collected again and will include the NPRS, global rating of changes (GROC), cervical range of motion, and DCF. The therapist will determine the next appropriate follow-up visit. Data will again be collected at the beginning of the 2nd visit follow-up and will include NPRS, GROC, cervical range of motion, DCF, PSFS, and NDI by the blinded physical therapist. Treatments of cervical and thoracic mobilization or manipulation will occur again based on group allocation established prior. The technique used by the treating clinician will be based on their assessment of the patient and again will follow group allocation. After the 2nd visit (day 3), the treating physical therapist is able to add or remove treatments, as they deem necessary to improve the patient's condition. Orthopedic manual therapy (mobilization or manipulation) may be adjusted based on patient need as well. Subsequent visits and plan of care will continue under the direction of the physical therapist based on the patient's need. Final data collection performed at discharge will include the NDI, PSFS, GROC, and total number of visits, patient satisfaction, therapist equipoise, and total days of care.

Analysis: Baseline characteristics of all subjects will be compared using either a t-test or chi square as appropriate. A two way multivariate analysis of variance (MANOVA) will be used to compare outcomes of NDI, PSFS, and NPRS at baseline, at day 3, and at day 30.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18-70 years old with a chief complaint of reproducible neck pain and an NDI score of 10 or greater.

Exclusion Criteria:

* Subjects are excluded if they have had recent whiplash or significant trauma, demonstrate red flag items such as malignancy, radiculopathy, myelopathy, fracture, metabolic disease, rheumatoid arthritis, long-term steroid use, or history of neck surgery. Additional exclusion criteria including neck pain of <2 on the NPRS, PSFS ≤ 8, no prior treatment within 6 weeks time, upper limb symptoms, or any pending litigation. Finally, if a therapist determines the patient has a neck condition that is highly irritable where the manipulation is not appropriate, they will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) | Initial evaluation, 2nd visit expected average day 3, and discharge expected average 4 weeks.
  The NDI is a reliable and valid outcome tool for patients with neck pain. It is a self-report measurement tool that was specifically constructed to measure the degree of disability for persons with neck pain. There are 10 total items that are ranked from 0-5 giving a total possible number of 50 points. The larger the score, the greater the disability for that individual.

SECONDARY OUTCOMES:
change in numeric pain rating scale (NPRS) | initial evaluation, 2nd visit expected average day 3, discharge expected average 4 weeks
  The NPRS is used to determine the patient's pain level. The patient is asked to rate their level of pain on an 11-point numerical scale 0-10 with 0 being "no pain" and 10 being the "worst possible pain."
Change in patient specific functional scale (PSFS) | Initial evaluation, 2nd visit expected average day 3, and at discharge expected average 4 weeks.
  The PSFS is a three item questionnaire where the patient is asked to list 3 items they are having difficulty with and rate them on a 0-10 scale with 0 being unable to perform and 10 being able to perform with no limitation.
Change in the global rating of change | after visit 2 (expected average day 3) and again at discharge expected average 4 weeks.
  The global rating of change is a 15-point scale where 0 is no change in condition, -7 is a very great deal worse and +7 is a very great deal better. The patient is asked to rate their overall current current condition compared with when they first started care.
Percent recovery | Measured at discharge expected average of 4 weeks into protocol
  The patient is asked to rate their overall improvement on a scale of 0% (no better) to 100% completely better
Change in deep cervical flexor endurance test | Initial examination, after 2 visit (expected average day 3) and at discharge ( expected average 4 weeks),
  The patient lies in supine and maximally tucks chin to activate the deep cervical flexors. The patient then is asked to lift their head 0.5-1.0 inches off the table and maintain the chin tuck and hold for as long as possible. The investigator times the hold and records when the position cannot be maintained any longer.

CONTACTS AND LOCATIONS:
Overall Officials: David W. Griswold, DPT, Principal Investigator — Youngstown State University; David W Griswold, DPT, Principal Investigator — Youngstown State University
Locations (2):
- United States (2):
  - Rehabilitex Inc., Solon, Ohio
  - Pain Relief and Physical Therapy, Havertown, Pennsylvania

REFERENCES:
- [Result] Dunning JR, Cleland JA, Waldrop MA, Arnot CF, Young IA, Turner M, Sigurdsson G. Upper cervical and upper thoracic thrust manipulation versus nonthrust mobilization in patients with mechanical neck pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):5-18. doi: 10.2519/jospt.2012.3894. Epub 2011 Sep 30. PMID 21979312
- [Result] Cross KM, Kuenze C, Grindstaff TL, Hertel J. Thoracic spine thrust manipulation improves pain, range of motion, and self-reported function in patients with mechanical neck pain: a systematic review. J Orthop Sports Phys Ther. 2011 Sep;41(9):633-42. doi: 10.2519/jospt.2011.3670. Epub 2011 Aug 31. PMID 21885904
- [Result] Lau HM, Wing Chiu TT, Lam TH. The effectiveness of thoracic manipulation on patients with chronic mechanical neck pain - a randomized controlled trial. Man Ther. 2011 Apr;16(2):141-7. doi: 10.1016/j.math.2010.08.003. Epub 2010 Sep 1. PMID 20813577
- [Result] Leaver AM, Refshauge KM, Maher CG, Latimer J, Herbert RD, Jull G, McAuley JH. Efficacy of manipulation for non-specific neck pain of recent onset: design of a randomised controlled trial. BMC Musculoskelet Disord. 2007 Feb 26;8:18. doi: 10.1186/1471-2474-8-18. PMID 17324291
- [Result] Miller J, Gross A, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL. Manual therapy and exercise for neck pain: A systematic review. Man Ther. 2010 Jun 1. doi: 10.1016/j.math.2010.02.007. Online ahead of print. PMID 20627797